CLINICAL TRIAL: NCT05726981
Title: Ultrasound and Cytological Evaluation 3 Years After Radiofrequency Thermal Ablation of Benign Thyroid Nodules : a Prospective Exploratory Cohort of 180 Nodules
Acronym: CYTOTHYRAF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP211436
Record Dates: First submitted 2023-01-12; First posted 2023-02-14 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Thermal Ablation; Fine Needle Aspiration Biopsy; Thyroid Nodules
MeSH Terms: conditions — Thyroid Nodule | interventions — Biopsy, Fine-Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with nodules treated by thermal ablation (Experimental): The study population is a monocentric cohort of patients who underwent thermoablation treatment for benign thyroid nodules 3 years ago. These patients aged >18 years-old were carriers of a benign but troublesome thyroid nodule before thermal ablation, either unique or "dominant", i.e. associated with one or more other non-significant nodules (<20 mm) that were subjected to simple ultrasound surveillance. Patients refused, after clear and fair information, surgical management of their nodule. On average, 2 patients have been treated for TA per week in the Thyroid Disease and Endocrine Tumor Department since 2016. Patients systematically benefit from annual clinical and ultrasound monitoring as part of their follow-up in our Department.
  Interventions: Procedure: Fine needle aspiration biopsy (FNAB)

INTERVENTIONS:
Procedure: Fine needle aspiration biopsy (FNAB) — Thyroid FNAB is a minimally invasive procedure performed routinely by an experienced sonographer.
  It is a safe and brief procedure, performed with a 27G or 25G (very fine) needle (3 needles, i.e. 1 needle per pass)

SUMMARY:
There is no scientific data on post-thermal ablation cytological aspects, but treated nodules that grow back significantly after a procedure justify a new cytology in order not to ignore a neoplastic process.

The EU-TIRADS classification usually used to stratify the risk of cancer (and to justify a fine needle aspiration biopsy) of thyroid nodules is not validated for nodules treated by thermal ablation (TA) (post-RF nodules). However, these nodules often acquire ultrasound criteria of suspicion making it necessary to develop an ultrasound stratification of the risk of malignancy specific to nodules treated by TA.

The objective of this work is to describe the ultrasound and cytological aspects of these treated nodules by performing a systematic assessment at 3 years after thermal ablation including systematic neck ultrasound and fine needle aspiration biopsy. Thus, an ultrasound and cytological atlas (Bethesda classification 2017) of nodules treated by thermal ablation will be constituted.

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 18 years old
2. Carrier of a benign thyroid nodule that has undergone radiofrequency thermoablation 36 months previously ± 12 months +/- 1 month, whether the nodule is stable, progressing or decreasing in volume during the screening period and/or on the day of inclusion.
3. Obtaining written informed consent
4. Affiliation to a social security system (excluding AME)

Exclusion Criteria:

1. Pregnant or breastfeeding women
2. Previous alcohol use
3. Patients on anti-vitamin K anticoagulants
4. Patients on direct oral anticoagulants
5. Persons deprived of liberty by judicial or administrative decision
6. Persons under forced psychiatric care
7. Persons admitted to a health or social institution for purposes other than research
8. Persons of full age who are under legal protection (guardianship or curatorship)
9. Persons unable to express their consent
10. Persons under a legal protection measure (there can be no derogation for this category)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-06-29 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Cytological change after thermoablation, as described by the 2017 Bethesda classification in six classes, scale ranging from I to VI. | Day of the Fine Needle Aspiration Biopsy
  Cytological result of the nodule 3 years after thermoablation, the result of which is given according to the 2017 Bethesda classification in six classes ranging from I to VI.

SECONDARY OUTCOMES:
Ultrasound description of the nodule: size (length x width x thickness) | Day of the Fine Needle Aspiration Biopsy
Ultrasound description of the nodule: volume (length x width x thickness) | Day of the Fine Needle Aspiration Biopsy
Ultrasound description of the nodule: echogenicity, as compared with the adjacent thyroid and muscular tissues | Day of the Fine Needle Aspiration Biopsy
Ultrasound description of the nodule: echostructure, measured as the percentage of liquid volume compared to nodule's total volume | Day of the Fine Needle Aspiration Biopsy

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Pitié-Salpêtrière - Department of Thyroid and Endocrine Tumour Pathologies, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided